CLINICAL TRIAL: NCT02543502
Title: Treatment of Periodontal Disease in Patients With Acute Myocardial Infarction: Randomized Controlled Trial
Brief Title: Treatment of Periodontal Disease in Patients With Acute Myocardial Infarction
Acronym: TPAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP nº 4742. 12
Record Dates: First submitted 2015-08-27; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Periodontitis
Keywords: Periodontitis; atherosclerosis; Heart Disease
MeSH Terms: conditions — Periodontitis; Atherosclerosis; Heart Diseases | interventions — Periodontal Index

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- periodontal treatment (Experimental): Group will receive treatment: periodontal treatment
  Interventions: Procedure: periodontal treatment
- Control Group. (No Intervention): Group will not receive treatment: periodontal treatment

INTERVENTIONS:
Procedure: periodontal treatment — treatment of periodontal cleaning
  Arms: periodontal treatment

SUMMARY:
The main objective of this study is to evaluate the effect of treatment periodontal endothelium-dependent artery of the arm in patients with acute myocardial infarction with ST-segment elevation undergoing primary coronary intervention.

DETAILED DESCRIPTION:
The present work sample will be composed by individuals who suffered from ST segment elevation myocardial infarction admitted to the Cardiologic Institute from Porto Alegre. Participants period of selection and evaluation extended from August 20th, 2012 to January 2015. The whole selection was performed by the responsible researcher, assessing periodontal condition of the individuals in the hospital bed. The participants will be accompanied during the hospital stay and outpatient basis, an expected average of six months.

Clinical Exam

Patients selected for the test group will receive periodontal examination in private offices. For the clinical exam, odontoscopy (Duflex®, Brasil) and Flórida 10mm periodontal catheters measured in millimeters (Newmar®, Brasil) will be employed. The clinical exam will be performed by an experienced periodontist (the same one who will perform the patients' treatment) and will include the evaluation of parameters related to the periodontal disease, which were noted by an assistant, in a standard form (Attachment A). All permanent teeth will be examined, except for the third molars. Periodontal variables will be evaluated in four sites per tooth (vestibular, distal, lingual and mesial), according to the following:

* Visible plaque index (VPI) - dental surfaces will be assessed by the naked eye after compressed air drying. Codes: 0 = absence of visible plaque, and 1 = presence of visible plaque (AINAMO and BAY, 1975).
* Catheterization Depth (CD) - distance from the gingival edge to the most apical portion able to be catheterized, in millimeters.
* Bleeding during Catheterization (BC): It will be registered the presence (score 1) or absence (score 0) of bleeding 30 seconds after measuring the catheterization depth
* Loss of Insertion (LI): It will be calculated through the distance between the amelocemental junction to the most apical portion of the periodontal pocket. This measurement will be performed in millimeters and always rounded down to the lowest mark.

Endothelial Function Exam Endothelial function assessment will be performed through endothelial dependent dilation of the brachial artery, observed through ultrasound with a linear 3-12 MHz transducer (EnVisor CHD, Philips, Bothell, WA, USA). Automated measurements of the vase diameter will be performed with a software from the equipment used in the procedure. The evaluations will be performed in the morning period, after an 8-hour fast, in controlled temperature (22°C). After ten minutes of rest, the images of the brachial artery will be recorded with a linear transducer continuously placed over the antecubital fossa for one minute (basal). The sphygmomanometer will be placed in the arm and insufflated to the edge of 50mmHG above systolic arterial pressure for five minutes, and the alteration in the diameter of the brachial artery 60 seconds after the cuff deflation will be compared to the basal diameter. The images of the vase in the end of the diastole (identified by the R wave in the ECG) will be digitalized and recorded in 3 second gaps during the whole procedure, being subsequently analyzed offline, using the software of the equipment used in the procedure.

After 10 minutes of rest, new measurements will be performed, measuring the endothelial dependent dilation through the administration of 25mg sublingual nytroglycerin. The flow measuring will be performed with a Doppler wave pulse at an angle of 70o. The increase in the blood flow after the arterial pressure liberation from the cuff will be expressed as reflex hyperemia (value for reflex hyperemia, divided by the baseline value for blood flow in the forearm). After one hundred and eighty days (6 months) a new Endothelial function assessment will be performed.

Periodontal Treatment Periodontal treatment will be performed by an expert in periodontics, in a private office, in the following treatment order. First, the case will be presented to the patients, providing information about periodontal diseases etiopathogeny, focusing on the importance of bacterial supragingival biofilm control for the treatment success. Afterwards, all the plaque retentive factors (dental calculus) will be removed in a single session. Decay lesions will be restored with provisional material; radicular debris will be extracted, and badly adapted restoration will be adjusted. Supragingival calculus will be removed with periodontal Gracey curettes (Newmar®, São Paulo, Brasil), followed by supragingival smoothing and polishing with rubber cup, prophylactic paste, dental floss and/or interdental brush. In the same session, participants will receive instructions on personalized oral hygiene, with multibristle brushes, toothpaste, dental floss and interdental brushes.

Fourteen days after the first appointment, under gingival radicular scraping and smoothing will be initiated (UGSS) with periodontal files and curettes (Newmar®, São Paulo, Brasil), under local anaesthesia, for a maximum period of four weeks. By the end of each UGSS appointment, patients will receive professional plaque removal and oral hygiene reinforcement, according to individual needs, for motivation and effective behavior change regarding to oral health care.

After periodontal treatment, patients from the test group will receive clinical reassessment after ninety days for hygiene reinforcement and professional teeth plaque removal. After one hundred and eighty days (6 months) a new complete periodontal exam will be performed.

Sample Calculation Minimum sample size will be calculated in 88 patients to detect a flow mediated dilation difference of 1% between the two study groups, with an average standard deviation of 1,67%, for a p<0,05 and statistical power of 90%.

Randomization Patients will be selected and invited to participate during hospital admission. Randomization will be performed two weeks after hospital discharge. Patients will be randomly distributed through the use of a computer generated table (randomization.com), to receive periodontal treatment (test group) or to participate in the control group, which will not receive any clinical intervention during the experiment period, but will be referred to periodontal treatment after the experimental period.

Blinding Endothelial disfunction evaluation will be performed by a professional that won't be aware of group allocation of each patient (test or control), either in the begging or end of the study.

Statistical Analysis Data will be presented as means and standard deviation, with confidence intervals of 95%, and relative and absolute frequencies. All the analysis will be based on the intention to treat principle. t Student test for impaired samples will be used to compare periodontal exam values before and after treatment. General estimative equations method, followed by multiple comparisons with bonferroni correction will be used to compare the DMF percentage intra and intergroup (intervention x control), and the covariance analysis will be used to compare the DMF variation (before and after treatment delta) between the control and intervention group, adjusted to the initial values. All data will be analyzed by SPSS software, version 22, and the significance value considered in the analysis of 0,05.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to our institution with a diagnosis of AMI (ST segment elevation> 0.1mV)
* older than 30 years
* with more than 8 teeth in the mouth
* with advanced periodontal disease

Exclusion Criteria:

* acute or chronical infection
* impossibility of attending the following interviews and/or the periodontal treatment
* refusing to signing the consent form
* individuals with substance abuse
* anticonvulsants and immunosuppressant drugs users
* pregnant and \ or lactating women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The difference in dilation measured by brachial artery blood flow | 6 months
  The primary outcome will be the difference in the dilation measured through the flow in the brachial artery by the end of six months.

SECONDARY OUTCOMES:
Major cardiovascular events | 6 months
  . The secondary outcomes will be major cardiovascular events (death, re-AMI, new revascularization and readmission for cardiovascular causes).

OTHER OUTCOMES:
Bacteremia | 24 hours
  ). Safe outcomes will be the occurence of bacteremia and/or excessive gingival bleeding during the procedure or within the following 24 hours. Bacteremia will be defined by the presence of fever and shivering with positive blood culture. Gingival bleeding will be evaluated by the gingival bleeding index.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Sc Quadros, Phd, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul, IC-FUC
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Schmidt MI, Duncan BB, Azevedo e Silva G, Menezes AM, Monteiro CA, Barreto SM, Chor D, Menezes PR. Chronic non-communicable diseases in Brazil: burden and current challenges. Lancet. 2011 Jun 4;377(9781):1949-61. doi: 10.1016/S0140-6736(11)60135-9. Epub 2011 May 9. PMID 21561658
- [Background] Bahekar AA, Singh S, Saha S, Molnar J, Arora R. The prevalence and incidence of coronary heart disease is significantly increased in periodontitis: a meta-analysis. Am Heart J. 2007 Nov;154(5):830-7. doi: 10.1016/j.ahj.2007.06.037. Epub 2007 Aug 20. PMID 17967586
- [Background] D'Aiuto F, Parkar M, Tonetti MS. Acute effects of periodontal therapy on bio-markers of vascular health. J Clin Periodontol. 2007 Feb;34(2):124-9. doi: 10.1111/j.1600-051X.2006.01037.x. Epub 2007 Jan 3. PMID 17214734
- [Background] Humphrey LL, Fu R, Buckley DI, Freeman M, Helfand M. Periodontal disease and coronary heart disease incidence: a systematic review and meta-analysis. J Gen Intern Med. 2008 Dec;23(12):2079-86. doi: 10.1007/s11606-008-0787-6. Epub 2008 Sep 20. PMID 18807098
- [Background] Libby P, Ridker PM, Hansson GK; Leducq Transatlantic Network on Atherothrombosis. Inflammation in atherosclerosis: from pathophysiology to practice. J Am Coll Cardiol. 2009 Dec 1;54(23):2129-38. doi: 10.1016/j.jacc.2009.09.009. PMID 19942084
- [Background] Lockhart PB, Bolger AF, Papapanou PN, Osinbowale O, Trevisan M, Levison ME, Taubert KA, Newburger JW, Gornik HL, Gewitz MH, Wilson WR, Smith SC Jr, Baddour LM; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee of the Council on Cardiovascular Disease in the Young, Council on Epidemiology and Prevention, Council on Peripheral Vascular Disease, and Council on Clinical Cardiology. Periodontal disease and atherosclerotic vascular disease: does the evidence support an independent association?: a scientific statement from the American Heart Association. Circulation. 2012 May 22;125(20):2520-44. doi: 10.1161/CIR.0b013e31825719f3. Epub 2012 Apr 18. PMID 22514251
- [Background] Ridker PM. C-reactive protein, inflammation, and cardiovascular disease: clinical update. Tex Heart Inst J. 2005;32(3):384-6. No abstract available. PMID 16392225
- [Background] Tonetti MS, D'Aiuto F, Nibali L, Donald A, Storry C, Parkar M, Suvan J, Hingorani AD, Vallance P, Deanfield J. Treatment of periodontitis and endothelial function. N Engl J Med. 2007 Mar 1;356(9):911-20. doi: 10.1056/NEJMoa063186. PMID 17329698
- [Background] Yu YH, Chasman DI, Buring JE, Rose L, Ridker PM. Cardiovascular risks associated with incident and prevalent periodontal disease. J Clin Periodontol. 2015 Jan;42(1):21-8. doi: 10.1111/jcpe.12335. Epub 2015 Jan 9. PMID 25385537
- [Background] Albandar JM, Brunelle JA, Kingman A. Destructive periodontal disease in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):13-29. doi: 10.1902/jop.1999.70.1.13. PMID 10052767
- [Background] Castro GD, Oppermann RV, Haas AN, Winter R, Alchieri JC. Association between psychosocial factors and periodontitis: a case-control study. J Clin Periodontol. 2006 Feb;33(2):109-14. doi: 10.1111/j.1600-051X.2005.00878.x. PMID 16441734
- [Background] D'Aiuto F, Parkar M, Andreou G, Suvan J, Brett PM, Ready D, Tonetti MS. Periodontitis and systemic inflammation: control of the local infection is associated with a reduction in serum inflammatory markers. J Dent Res. 2004 Feb;83(2):156-60. doi: 10.1177/154405910408300214. PMID 14742655
- [Background] D'Aiuto F, Parkar M, Tonetti MS. Periodontal therapy: a novel acute inflammatory model. Inflamm Res. 2005 Oct;54(10):412-4. doi: 10.1007/s00011-005-1375-4. PMID 16283108
- [Background] Elter JR, Hinderliter AL, Offenbacher S, Beck JD, Caughey M, Brodala N, Madianos PN. The effects of periodontal therapy on vascular endothelial function: a pilot trial. Am Heart J. 2006 Jan;151(1):47. doi: 10.1016/j.ahj.2005.10.002. PMID 16368290
- [Background] Joshipura KJ, Wand HC, Merchant AT, Rimm EB. Periodontal disease and biomarkers related to cardiovascular disease. J Dent Res. 2004 Feb;83(2):151-5. doi: 10.1177/154405910408300213. PMID 14742654
- [Background] Libby P, Okamoto Y, Rocha VZ, Folco E. Inflammation in atherosclerosis: transition from theory to practice. Circ J. 2010 Feb;74(2):213-20. doi: 10.1253/circj.cj-09-0706. Epub 2010 Jan 9. PMID 20065609
- [Background] Pussinen PJ, Tuomisto K, Jousilahti P, Havulinna AS, Sundvall J, Salomaa V. Endotoxemia, immune response to periodontal pathogens, and systemic inflammation associate with incident cardiovascular disease events. Arterioscler Thromb Vasc Biol. 2007 Jun;27(6):1433-9. doi: 10.1161/ATVBAHA.106.138743. Epub 2007 Mar 15. PMID 17363692
- [Background] Ramirez JH, Arce RM, Contreras A. Periodontal treatment effects on endothelial function and cardiovascular disease biomarkers in subjects with chronic periodontitis: protocol for a randomized clinical trial. Trials. 2011 Feb 16;12:46. doi: 10.1186/1745-6215-12-46. PMID 21324167
- [Background] Teeuw WJ, Slot DE, Susanto H, Gerdes VE, Abbas F, D'Aiuto F, Kastelein JJ, Loos BG. Treatment of periodontitis improves the atherosclerotic profile: a systematic review and meta-analysis. J Clin Periodontol. 2014 Jan;41(1):70-9. doi: 10.1111/jcpe.12171. Epub 2013 Oct 29. PMID 24111886
- [Background] Blum A, Front E, Peleg A. Periodontal care may improve systemic inflammation. Clin Invest Med. 2007;30(3):E114-7. doi: 10.25011/cim.v30i3.1079. PMID 17716549
- [Background] Pischon N, Hagewald S, Kunze M, Heng N, Christan C, Kleber BM, Muller C, Bernimoulin JP. Influence of periodontal therapy on the regulation of soluble cell adhesion molecule expression in aggressive periodontitis patients. J Periodontol. 2007 Apr;78(4):683-90. doi: 10.1902/jop.2007.060286. PMID 17397316
- [Background] Li X, Tse HF, Jin LJ. Novel endothelial biomarkers: implications for periodontal disease and CVD. J Dent Res. 2011 Sep;90(9):1062-9. doi: 10.1177/0022034510397194. Epub 2011 Feb 14. PMID 21321068
- [Background] Li X, Tse HF, Yiu KH, Li LS, Jin L. Effect of periodontal treatment on circulating CD34(+) cells and peripheral vascular endothelial function: a randomized controlled trial. J Clin Periodontol. 2011 Feb;38(2):148-56. doi: 10.1111/j.1600-051X.2010.01651.x. Epub 2010 Dec 6. PMID 21133981
- [Background] Piconi S, Trabattoni D, Luraghi C, Perilli E, Borelli M, Pacei M, Rizzardini G, Lattuada A, Bray DH, Catalano M, Sparaco A, Clerici M. Treatment of periodontal disease results in improvements in endothelial dysfunction and reduction of the carotid intima-media thickness. FASEB J. 2009 Apr;23(4):1196-204. doi: 10.1096/fj.08-119578. Epub 2008 Dec 12. PMID 19074511
- [Background] Amar S, Gokce N, Morgan S, Loukideli M, Van Dyke TE, Vita JA. Periodontal disease is associated with brachial artery endothelial dysfunction and systemic inflammation. Arterioscler Thromb Vasc Biol. 2003 Jul 1;23(7):1245-9. doi: 10.1161/01.ATV.0000078603.90302.4A. Epub 2003 May 22. PMID 12763762
- [Background] Mercanoglu F, Oflaz H, Oz O, Gokbuget AY, Genchellac H, Sezer M, Nisanci Y, Umman S. Endothelial dysfunction in patients with chronic periodontitis and its improvement after initial periodontal therapy. J Periodontol. 2004 Dec;75(12):1694-700. doi: 10.1902/jop.2004.75.12.1694. PMID 15732873
- [Background] Saffi MA, Furtado MV, Polanczyk CA, Montenegro MM, Ribeiro IW, Kampits C, Haas AN, Rosing CK, Rabelo-Silva ER. Relationship between vascular endothelium and periodontal disease in atherosclerotic lesions: Review article. World J Cardiol. 2015 Jan 26;7(1):26-30. doi: 10.4330/wjc.v7.i1.26. PMID 25632316
- [Background] Seinost G, Wimmer G, Skerget M, Thaller E, Brodmann M, Gasser R, Bratschko RO, Pilger E. Periodontal treatment improves endothelial dysfunction in patients with severe periodontitis. Am Heart J. 2005 Jun;149(6):1050-4. doi: 10.1016/j.ahj.2004.09.059. PMID 15976787
- [Derived] Lobo MG, Schmidt MM, Lopes RD, Dipp T, Feijo IP, Schmidt KES, Gazeta CA, Azeredo ML, Markoski M, Pellanda LC, Gottschall CAM, Quadros AS. Treating periodontal disease in patients with myocardial infarction: A randomized clinical trial. Eur J Intern Med. 2020 Jan;71:76-80. doi: 10.1016/j.ejim.2019.08.012. Epub 2019 Dec 4. PMID 31810741